CLINICAL TRIAL: NCT01771315
Title: Nurse Led Follow-up After Total Knee Arthroplasty - a Randomized Trial
Brief Title: Nurse Led Follow-up After Total Knee Arthroplasty
Acronym: NFTKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Birte Oestergaard, Associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UNR-2013112-4; R108-A2423 (Other Grant/Funding Number: The Danish Rheumatism Association)
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty; telephone follow-up; physical function; health related quality of life; self-efficacy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telephone follow-up (Experimental): Nurse led follow-up in form of consultation by telephone 4 days and 2weeks after discharge, respectively as a supplement to conventional admission course.
  Interventions: Behavioral: Telephone follow-up
- Usual treatment (No Intervention): All patients follow conventional admission course which implies preoperative seminar and a discharge planning consultation on the day of discharge. The patients are discharged to home, referred to physiotherapy in the community and a scheduled follow-up by the surgeon after 3 month in the orthopedic outpatient clinic.

INTERVENTIONS:
Behavioral: Telephone follow-up — The consultation is structured by predefined themes relevant for identifying health related problems in regard to illness to give adequate education and counseling. The form of each consultation will vary according to the individual needs of the patients.
  Arms: telephone follow-up

SUMMARY:
The aim of this study is to determine the effect of nurse led follow-up following total knee arthroplasty in regard to physical function, health related quality of life and self-efficacy.

DETAILED DESCRIPTION:
Due to shorter hospitalization the patients early have to be responsible for their own rehabilitation. However, the patients experience a variety of health related problems in the rehabilitations period following total knee arthroplasty and they have difficulties transferring health related information to their home settings. Nurse led follow-up in the early rehabilitation period might improve the health status of the patients by improving their knowledge and skills to handle health related problems. No studies found has investigated the effect of nurse led follow-up in form of telephone call following total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* primary first-time total knee arthroplasty due to osteoarthrosis
* followed conventional admission course and discharged ≤ 4 days after surgery
* understand and talk Danish
* signed informed consent

Exclusion Criteria:

* in terminal phase of another serious illness such as i.e. cancer with expected lifetime less than 6 months
* previous total hip replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in physical function assessed by ≥ 12 points in physical function score in the Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index | 3 days, 1, 3, 6 and 12 months post-surgery
  The WOMAC Index is disease specific measuring health status om three subscales: pain, stiffness and physical function

SECONDARY OUTCOMES:
Change in the pain and stiffness score in WOMAC Index | 3 days, 1, 3, 6 and 12 months post-surgery
Changes in all scores in the subscales in Medical Outcomes Study Short Form (SF-36) | 3 days, 1, 3, 6 and 12 months post-surgery
  A generic measure of health related quality of life
Change in the score in the General Self-Efficacy Scale | 3 days, 1, 3 and 6 months post-surgery
  An unidimensional measure of general self-efficacy.
Number of acute visits to the orthopedic outpatient clinic | 3 days, 1, 3, 6 anf 12 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Szöts, Principal Investigator — University Hospital Gentofte
Locations (1):
- University Hospital Gentofte, Hellerup, Gentofte, Denmark

REFERENCES:
- [Derived] Szots K, Konradsen H, Solgaard S, Ostergaard B. Telephone follow-up by nurse following total knee arthroplasty - protocol for a randomized clinical trial (NCT 01771315). BMC Nurs. 2014 May 21;13:14. doi: 10.1186/1472-6955-13-14. eCollection 2014. PMID 24872728